CLINICAL TRIAL: NCT03331380
Title: Technical Development of Cardiovascular Magnetic Resonance Imaging (CMR) Using a Low Specific Absorption Rate (SAR) Scanner System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 180011; 18-H-0011
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12-02

CONDITIONS: CAD
Keywords: 1.5 T CMR; Low SAR CMR; Gadolinium; Regadenoson; Adenosine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group A (Other): Group A includes 600 healthy adult volunteers of both sexes with-out known cardiovascular disease
  Interventions: Device: MRI scan - obj 1; Device: MRI scans - obj 2
- Group B (Other): Group B includes 500 adult subjects of both sexes with known sta-ble cardiovascular disease including adults with stable coronary artery disease after myocardial infarction; adults with heart failure and reduced left ventricular systolic function; adults with pulmonary artery hypertension; adults with congenital heart disease including cardiac shunts; adults with valvular heart disease including aortic stenosis, mitral regurgitation, and tricuspid regurgitation; and adults with metallic cardiovascular implants (such as coronary and peripheral artery stents) known to be safe for CMR at 1.5T
  Interventions: Device: MRI scans - obj 3
- Group C (Other): Group C includes 500 adult subjects of both sexes with known non-cardiovascular disease
  Interventions: Device: MRI scans - obj 4

INTERVENTIONS:
Device: MRI scan - obj 1 — For objective 1 (protocol optimization), healthy volunteers undergo imaging using an investigational low SAR CMR scanner for up to two hours, some without and some with administration of intravenous gadolinium based contrast agents (GBCAs).
  Arms: Group A
Device: MRI scans - obj 2 — For objective 2 (comparative scanning of normals), healthy volunteers undergo two CMR examinations on two different MRI scanners (investigational low SAR CMR and conventional 1.5T CMR), some without and some with administration of intravenous GBCA.
  Arms: Group A
Device: MRI scans - obj 3 — For objective 3 (comparative scanning of patients), subjects with known stable cardiovascular disease undergo two CMR examinations on two different MRI scanners (investigational low SAR CMR and conventional 1.5T CMR), some without and some with administration of intravenous GBCA.
  Arms: Group B
Device: MRI scans - obj 4 — For objective 4 (comparative scanning of patients), subjects with known or suspected disease, including neurological, musculoskeletal disease, abdominal or lung disease, will undergo two MR examinations on two different MRI scanners (investigational low SAR CMR and conventional MR).
  Arms: Group C

SUMMARY:
Background:

Researchers are testing version of a system known as a magnetic resonance imagining (MRI) scanner that uses strong magnetic fields, radio waves and the like to create images of the organs in the body. It uses lower energy levels than other MRI scanners. This may help scan people with metal devices in their body, or in invasive heart procedures using metal tools.

Objective:

To test a new MRI scanner and software changes to create better pictures.

Eligibility:

People with disease and healthy volunteers, ages 18 and older.

Design:

Participants will be screened with blood tests.

Participants may have both the new MRI and a conventional MRI or only the new one. If 2 are done, they must be within 60 days.

For both MRI versions, participants lie on a table that slides into a large tube. During scans, they will hold their breath for up to 20 seconds at a time. Heart activity will be measured by wires connected to pads on the skin. A flexible belt may be used to monitor their breathing. They will be in the scanner up to 2 hours.

Participants can agree to have a dye called gadolinium injected into their arm during the scan. This brightens the pictures.

Participants can agree to take a drug called a vasodilator. This helps detect areas of the heart with abnormal blood supply. Scans of the heart are taken before, during, and after they get the medicine. The drug may cause temporary chest pain or shortness of breath. They may get other drugs to relieve these symptoms.

Sponsoring Institution: National Heart, Lung, and Blood Institute

DETAILED DESCRIPTION:
Cardiac magnetic resonance imaging (CMR) provides accurate and reproducible measures of cardiac chamber volumes, cardiac function, blood flow, myocardial scar, myocardial extracellular volume as a measure of collagen content, myocardial iron content, and others, all without exposure to ionizing radiation. The prevailing wisdom is that CMR using high specific absorption rate (SAR) scanning modes produces highest image quality. We propose a method of CMR that can be performed with low SAR but that nevertheless preserves image quality because of efficient use of CMR signal. CMR using low SAR is attractive because it may reduce heating of metallic structures. This may allow safe CMR in patients with metallic implants, and it may allow MRI catheterization using metallic guidewires and catheter devices.

The goal of this non-significant risk (NSR) medical device study is to test initial technical feasibility of low SAR CMR in healthy volunteers by technical optimization of scanner protocols, to test comparative accuracy of standard CMR measurements in healthy volunteers using low SAR CMR versus conventional CMR, and to test comparative accuracy of standard CMR measurements in adult patients with known stable heart disease using low SAR CMR versus conventional CMR. A secondary goal is to assess the potential of this new low SAR CMR system to perform non-cardiovascular radiological diagnostic imaging by testing comparative diagnostic accuracy of standard MR measurements in adult patients with known non-cardiovascular disease using the low SAR CMR system vs conventional MR exam.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for All Participants (Objectives 1, 2, 3, and 4)

* Men and women age greater than or equal to 18 years
* Able to provide informed consent in writing
* Willingness to cooperate with all study procedures (including food restriction) and available for scheduled study events

Inclusion Criteria for Healthy Volunteers (Objectives 1 and 2)

-Currently healthy, self-reported

Inclusion Criteria for Subjects with Heart Disease (Objective 3)

* Subjects having known heart disease including but not limited to
* Stable angina pectoris due to epicardial coronary artery obstruction
* Past myocardial infarction
* Heart failure with reduced ejection fraction
* Valvular heart disease
* Pulmonary artery hypertension
* Congenital heart disease with or without prior repair
* Myocarditis
* Infiltrative cardiomyopathy
* Hypertrophic cardiomyopathy

Inclusion Criteria for Subjects with Non-Cardiac Disease (Objective 4)

* Having known brain disease including but not limited to:

  * Transient ischemic attack or stroke after 24 hours of onset
  * Infection, inflammation meningitis
  * Cognitive decline, neurodegenerative disorders
  * Demyelinating disease, multiple sclerosis
  * Loss of consciousness, seizures, epilepsy
  * Brain tumor, metastases, abscess, lesion
  * Vascular pathology
  * Headache
  * Hemorrhage
  * Trauma
* Have known musculoskeletal disease including but not limited to:

  * Persistent neck pain or radiculopathy
  * Cancer or tumors of the spine
  * Congenital abnormalities of the spinal cord or knee
  * Multiple sclerosis
  * Injury or trauma
  * Fracture evaluation
  * Infectious or inflammatory processes
  * Soft tissue damage
  * Muscle or tendon disorders
  * Knee meniscal disorders
  * Marrow abnormalities
  * Mechanical knee symptoms
  * Vascular conditions
* Have known abdominal diseases including but not limited to:

  * Bowel obstruction
  * Masses and tumors
  * Crohns disease
  * Diffuse liver disease such as hemochromatosis, hemosiderosis, fatty infiltration
  * Focal hepatic lesions
  * Cirrhotic liver
  * Iron content determination
  * Cystic kidney disease
  * Vascular abnormalities
* Have known lung disease including but not limited to:

  * Cancer, tumors and masses
  * Vascular and lymphatic abnormalities
  * Pulmonary thromboembolic disease
  * Trauma
  * Suspected bronchiolitis
  * Bronchiectasis or pneumonitis
  * Asthma and other obstructive lung diseases
  * Pulmonary lymphangioleiomyomatosis
  * Cystic and interstitial lung diseases such as pulmonary lymphangioleiomyomatosis and cystic fibrosis
* Have other known non-cardiovascular disease

Inclusion criteria for bronchodilators:

- Only subjects who use bronchodilators routinely or those have undergone previous pulmonary function testing with bronchodilators will be invited to undergo bronchodilator testing during MRI.

EXCLUSION CRITERIA:

Exclusion Criteria for All Participants:

* Conditions that are thought to make MRI unsafe (that will be determined by filling out a separate form) including:

  * Cerebral aneurysm clip unless it is labeled safe for MRI
  * Neural stimulator (e.g. TENS-Unit) unless it is labeled safe for MRI
  * Any type of ear implant unless it is labeled safe for MRI
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe for MRI
* Pregnancy. When uncertain, subjects will undergo either urine or serum pregnancy testing. Results from up to 3 days prior to the examination will be used. Post-menopausal and surgically sterilized subjects are exempt from this testing.

  * If a urine or serum pregnancy test was administered as part of a referral protocol, and the test was administered up to 3 days prior to MRI examination for this protocol, a new pregnancy test will not be required for this protocol.
  * If a pregnancy test has not been administered within 3 days of MRI examination for this protocol, a serum or urine pregnancy test will be administered. Medical personnel will determine which pregnancy test is appropriate based on subject s medical history, screening, and individual scenario. In addition, the subject will be asked if she may be pregnant prior to the performance of the MRI, even if the pregnancy test was negative within the past week. The pregnancy test will be repeated if she answers in the affirmative.

Exclusion Criteria for Gadolinium:

-When gadolinium based contrast agent (GBCA) exposure is planned

* Objective 1 and 2, Healthy Volunteers: No gadolinium based contrast agent exposure is permitted if eGFR < 60 mL/min/1.73m^(2) using the CKD-EPI equation or equivalent and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications.
* Objective 3 and 4, Volunteers with Cardiac and Non-Cardiac Disease: No gadolinium based contrast agent exposure is permitted if eGFR < 30 mL/min/1.73m^(2) using the CKDEPI equation [25] or equivalent and a serum creatinine measured within 2 weeks without

intercurrent change in medical condition or medications.

--For all objectives not more than two research MRI exams with GBCA exposure in a 12 month period. Research MRI exams performed outside of this protocol will be included in the 12 month period.

* Subjects meeting this exclusion criterion, or without eGFR determination, may still be included in the study but may not be exposed to gadolinium-based contrast agents
* Breast feeding (unless subject is willing to discard breast milk for 24 hours)
* Does not wish to be exposed to gadolinium.

Exclusion Criteria for Oxygen Inhalation:

* Severe chronic obstructive pulmonary disease defined as requiring more than one bronchodilator medication every day or continuous oxygen requiring
* Prior treatment with bleomycin

Exclusion Criteria for Ferumoxytol Contrast

* A history of allergic reaction to any intravenous iron product
* Allergy to ferumoxytol or to mannitol excipient
* Breast feeding
* Does not wish to be exposed to ferumoxytol
* Iron overload

Exclusion Criteria for oral contrast agent:

* A history of reaction to oral contrast (if using barium sulfate)
* Breast feeding unless subject is willing to discard breast milk for 24 hours (if using barium sulfate)
* Allergy to pineapple (if using pineapple juice)
* Does not wish to be exposed to oral contrast

Exclusion Criteria for Healthy Volunteers (Objectives 1 and 2)

-Important past medical illness

Exclusion Criteria for Adults with heart Disease (Objective 3)

* Unstable angina, acute coronary syndrome, or myocardial infarction not attributable to PCI, within 2 weeks unless after coronary revascularization of the culprit lesion.
* Any hemodynamic instability or decompensated heart failure as determined by the enrolling physician.
* Adenosine: Patients with asthma or chronic obstructive pulmonary disease of any severity are ineligible for vasodilator stress CMR with adenosine.
* Regadenoson: Only patients with severe or uncontrolled asthma or severe or uncontrolled chronic obstructive pulmonary disease are ineligible for vasodilator stress CMR with regadenoson. This will be determined at the discretion of the supervising provider based on medical records and physical exam.
* Patients with advanced heart block on baseline ECG are ineligible for vasodilator stress CMR

Exclusion Criteria for Adults with Non-Cardiac Disease (Objective 4)

* Acute illness for which investigational imaging might delay care (such as acute stroke before treatment), as determined by the enrolling physician
* Any hemodynamic instability as determined by the enrolling physician.

Exclusion criteria for bronchodilators:

- Patient refuses bronchodilator administration.

Exclusion criteria for adults with cardiac implanted electronic devices (CIED, pacemakers or defibrillators:

Low-SAR MRI:

* Subjects with MRI-conditional and legacy CIEDs are not excluded, based on the intrinsic safety of low-SAR MRI.
* Subjects with CIEDs are excluded if they have pacemakers implanted before 1998; ICDs implanted before 2000; temporary, epicardial or abandoned leads; and CIEDs implanted <4 weeks prior to MRI exam.

Conventional MRI:

-Subjects with CIED are excluded from conventional MRI unless they have CIEDs that are labeled as MRI conditional or MRI safe, and that are implanted greater than or equal to 4 weeks prior to MRI.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2950 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility and Non-inferiority of the above measurements and examinations ob-tained using low SAR CMR versus commercial CMR in healthy volun-teers and in patients with heart disease | 72 months
  To determine whether the the low SAR CMR is a feasible alternative to standard CMR

SECONDARY OUTCOMES:
Numerous exploratory secondary endpoints are sought around the listed measurements across MRI systems and disease states | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne E Campbell, Ph.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Xiang J, Ramasawmy R, Seemann F, Peters DC, Campbell-Washburn AE. Balanced steady-state free precession phase contrast at 0.55T applied to aortic flow. J Cardiovasc Magn Reson. 2024 Winter;26(2):101098. doi: 10.1016/j.jocmr.2024.101098. Epub 2024 Sep 13. PMID 39278416
- [Derived] Campbell-Washburn AE, Jiang Y, Korzdorfer G, Nittka M, Griswold MA. Feasibility of MR fingerprinting using a high-performance 0.55 T MRI system. Magn Reson Imaging. 2021 Sep;81:88-93. doi: 10.1016/j.mri.2021.06.002. Epub 2021 Jun 8. PMID 34116134
- [Derived] Bandettini WP, Shanbhag SM, Mancini C, Henry JL, Lowery M, Chen MY, Xue H, Kellman P, Campbell-Washburn AE. Evaluation of Myocardial Infarction by Cardiovascular Magnetic Resonance at 0.55-T Compared to 1.5-T. JACC Cardiovasc Imaging. 2021 Sep;14(9):1866-1868. doi: 10.1016/j.jcmg.2021.02.024. Epub 2021 May 19. No abstract available. PMID 34023254
- [Derived] Bandettini WP, Shanbhag SM, Mancini C, McGuirt DR, Kellman P, Xue H, Henry JL, Lowery M, Thein SL, Chen MY, Campbell-Washburn AE. A comparison of cine CMR imaging at 0.55 T and 1.5 T. J Cardiovasc Magn Reson. 2020 May 18;22(1):37. doi: 10.1186/s12968-020-00618-y. PMID 32423456
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0011.html